CLINICAL TRIAL: NCT03125681
Title: Effect of Remote Ischemic Conditioning on Platelet Dysfunction Following Off-pump Coronary Artery Bypass Surgery
Brief Title: Remote Ischemic Conditioning and Platelet Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIPC_multiplate
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Platelet Function
Keywords: remote ischemic conditioning; off-pump coronary artery bypass surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): Applying pneumatic cuff on upper extremity (5 minutes cycles of limb ischemia and reperfusion with pneumatic cuff up to 200 mmHg repeated by four times) before and after coronary anastomoses.
  Interventions: Procedure: Remote ischemic conditioning
- Control (Placebo Comparator): All the procedures were the same in the control group, except for the fact that the three-way stopcock between the pneumatic cuff and the cuff inflator was opened and therefore the cuff pressure did not increase.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote ischemic conditioning — In the RIC group, RIC is performed before and after coronary anastomoses by 5 minutes limb ischemia and reperfusion with pneumatic cuff up to 200 mmHg repeated by four times.
  Arms: Remote ischemic conditioning
Procedure: Control — In the control group, all the procedures will be same with RIC group, except for the fact that the three-way stopcock between the pneumatic cuff and the cuff inflator was opened and therefore the cuff pressure did not increase.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of remote ischemic conditioning on platelet function during off-pump coronary artery bypass surgery.

DETAILED DESCRIPTION:
Remote ischemic conditioning (RIC) may affect platelet function. However, little is known about effect of RIC on platelet function during off-pump coronary artery bypass surgery. In this study investigators are going to perform RIC after anesthesia induction (remote ischemic pre-conditioning) and after completion of coronary anastomoses (remote ischemic post-conditioning), and compare platelet function parameters with control group.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 80 years of adult patient undergoing elective off-pump coronary artery bypass surgery

Exclusion Criteria:

* Acute Myocardial Infarction
* Recent (<1 month) coronary angioplasty (percutaneous coronary intervention, PCI)
* Acute cerebrovascular ischemia (<6 months)
* Preoperative LV EF < 30%, mechanical ventricular support (IABP, VAD, ECMO)
* Peripheral vascular disease
* Poorly controlled diabetes mellitus
* Alzheimer's disease
* NSAIDs within 3 days
* iv heparin within 6 h
* low molecular weight heparin within 24 h
* platelet inhibitor within 24 h
* known thrombocytopenia
* renal failure / hemodialysis
* active infection
* preoperative bleeding diathesis
* redo-operation
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
Change of Multiplate ADPtest AUC | Baseline, at the end of surgery, postoperative day 1
  Area under the aggregation curve (AUC) after platelet stimulation with adenosine diphosphate

SECONDARY OUTCOMES:
Change of Multiplate ASPItest AUC | Baseline, at the end of surgery, postoperative day 1
  Area under the aggregation curve (AUC) after platelet stimulation with arachidonic acid
Change of Multiplate COLtest AUC | Baseline, at the end of surgery, postoperative day 1
  Area under the aggregation curve (AUC) after platelet stimulation with collagen
Change of Rotational thromboelastometry EXTEM parameter | Baseline, at the end of surgery, postoperative day 1
  Screening test for the extrinsic haemostasis system
Change of Rotational thromboelastometry FIBTEM parameter | Baseline, at the end of surgery, postoperative day 1
  Represents an EXTEM based assay for the fibrin part of the clot
Rotational thromboelastometry INTEM parameter | Baseline, at the end of surgery, postoperative day 1
  Intrinsically activated rotational thrombelastometry
Change of Rotational thromboelastometry HEPTEM parameter | Baseline, at the end of surgery, postoperative day 1
  Represents an INTEM assay performed in the presence of heparinase
Amount of peri-operative bleeding and transfusion | At the end of surgery, postoperative day 1,2,3
  Amount of peri-operative bleeding and transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, M.D., Ph. D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No